CLINICAL TRIAL: NCT04215354
Title: Association Between Fatigue and Balance in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Abeer Saeed Alawami, Master student, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2014-04-319
Record Dates: First submitted 2019-12-15; First posted 2020-01-02 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis
Keywords: MULTIPLE SCLEROSIS; FATIGUE; BALANCE
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Potential participants were informed that they will be randomly allocated in one of the three study groups: the magnet (BEMER) group, virtual reality (Wii) group or the placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MAGNET GROUP (Experimental): Patients were exposed to very low pulsed electromagnetic field induced by BEMER machine model type: B.BOX Professional using magnet mattress.
  Interventions: Device: Magnetic field
- VIRTUAL REALITY (Experimental): Balance training was done using the Wii Fit plus machine which required balance board .Using video game console designed by Nintendo.
  The program consisted of three games: soccer heading, ski slalom and table tilt.
  Interventions: Device: Virtual reality
- PLACEBO (Active Comparator): Patients in the placebo group had identical program to magnet group. They were asked to lie down in the magnet mattress; however, the magnet was not switched on and the patient doesn't know (blind).
  Interventions: Device: Magnetic field
- HEALTHY SUBJECT (No Intervention): healthy subjects with age, gender and BMI matched with the patients with MS were recruited to participate in the study. This group was recruited to establish the normal balance and fatigue parameters. Subjects in this group sign the consent form of healthy subjects and all measurement was taken as balance, fatigue, depression, quality of life and urinary incontinence screening questionnaire.

INTERVENTIONS:
Device: Magnetic field — Low pulsed electromagnetic field induced by BEMER machine model type: B.BOX Professional, model NO: 420200, 12-15 Volt, with maximum 300 Watt and average flux density around 35 microtesla- (BEMER Liechtenstein product, USA). Mattress which is flexible, 6 flat coil was used for whole body therapy.
  Other Names: BEMER
  Arms: MAGNET GROUP; PLACEBO
Device: Virtual reality — Wii Fit plus machine which required balance board . It is a video game console designed by Nintendo 2009
  Other Names: Wii
  Arms: VIRTUAL REALITY

SUMMARY:
The relationship between fatigue and balance was established. Fatigue was correlated with 8 parameters of balance scales. Moreover, there was a strong correlation between the level of fatigue from one side and depression, quality of life and disease severity from the other side.Fatigue seems to be the main problem in patients with MS which may influence other signs and symptoms such as balance.

DETAILED DESCRIPTION:
Electromagnetic field significantly reduced fatigue level in patients with MS.This effect reflected significantly on other symptoms such as balance, depression, disease severity and the quality of life in those patients.

Virtual reality program significantly improving balance and balance perception .Virtual reality program also improved quality of life by improving general health, physical function and decreasing physical limitation significantly. However, Virtual reality programs did not improve fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting type of MS.
* Age between 20-50 years.
* Ambulatory with or without an device.
* Complaining of fatigue, Have a score of 4/10 or more on the fatigue visual analogue scale in last four weeks

Exclusion Criteria:

* An acute episode of MS within the last 30 days.
* Pregnancy at any stage.
* Severely blurred vision.
* A pacemaker.
* Epilepsy of any type.
* Recent organ transplant.
* Cardiac arrhythmia.
* Large aneurysm.
* Heavy psychosis.
* Otitis media in last 2 weeks.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale | 12 weeks.
  It is a 21 items standardized questionnaire. Each item has five levels of response (range from 0 - 4). The total score ranges from 0 (no impact of fatigue) better condition to 84 (maximum impact of fatigue)worse condition.
Balance | 12 weeks.
  Berg Balance Scale (BBS)range from 0(worse condition) to 56(better condition)
balance confidence | 12 weeks.
  Activities- specific Balance Confidence scale .it is 16 items ofvisual analogue scale from 0-100%.score from 0 minimum confidence (worse condition) to 1600 maximum score (better condition).
Depression (Beck depression inventory ii (BDI-II)) | 12 weeks.
  It is 21 questions with each item range from 0 (normal) to 3 (most severe) with a maximum score of 63 (worse condition).The total score of the scale was used to classify patients as follows: normal (1-10), mild mood disturbance (11-16), border line of depression (17-20), moderate depression (21-30), severe depression (31-40), extreme depression (over 40)
Static balance using posturography, | 12 weeks
  stability levels range from 1 to 10, with 10 being the most stable or least difficult to perform. Static balance was measured at three different levels of stability; high level 8, medium 5 and low level 2. These levels where chosen to test patient balance on varying degree of instability.Patient who was unable to do the test due to sever balance impairment was given a score of 5000 based on the manufacturer recommendations in the machine manual (maximum score can subject got) which mean sever imbalance.

SECONDARY OUTCOMES:
Quality of life measurement (Short Form 36 (SF-36) | 12 weeks.
  The SF-36 consists of eight scaled scores as vitality (energy/fatigue), physical functioning, bodily pain, general health perceptions, and physical role functioning, emotional role functioning, social role functioning and mental health.each item is scored from 0-100 for total 1800. The lower the score the more the disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No